CLINICAL TRIAL: NCT02722798
Title: A Phase 2 Open-Label Trial to Assess the Efficacy and Safety of KRN23 in Patients With Tumor-Induced Osteomalacia or Epidermal Nevus Syndrome and a Post-marketing Study of KRN23 Switched From the Phase 2 Trial
Brief Title: A Study of KRN23 in Subjects With Tumor-Induced Osteomalacia or Epidermal Nevus Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-002
Record Dates: First submitted 2016-03-07; First posted 2016-03-30 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Tumor-Induced Osteomalacia or Epidermal Nevus Syndrome
MeSH Terms: conditions — Oncogenic osteomalacia; Nevus, Sebaceous of Jadassohn | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KRN23 (Experimental): Subjects will receive subcutaneous injections of KRN23 every 4 weeks from Week 0 through Week 224
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — Doses may be titrated to achieve the target peak serum phosphorus range

SUMMARY:
Before switching to the post-marketing study:

To evaluate the efficacy and safety of KRN23 after its 144-week once every 4 weeks (Q4W) repeated SC administration to Japanese and Korean patients with TIO or ENS by a multicenter, open-label, intraindividual dose adjustment study.

After switching to the post-marketing study:

To evaluate the safety and efficacy of KRN23, which is switched from the investigational product to the post-marketing investigational product, at the approved dose and dosing regimen in subjects who continue treatment after the marketing approval of KRN23 in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Diagnosis of Tumor-Induced Osteomalacia(TIO) or Epidermal Nevus Syndrome(ENS) and not amenable to receive surgical excision of the offending tumor/lesion
3. Serum phosphorus level < 2.5 mg/dL
4. Serum FGF23 level ≥ 100 pg/mL
5. Ratio of renal tubular maximum phosphate reabsorption rate to glomerular filtration rate< 2.5 mg/dL
6. Estimated glomerular filtration rate (eGFR) at screening ≥ 60 mL/min/1.73 m2, or eGFR ≥ 30 and < 60 mL/min/1.73 m2 with an evidence of no renal failure related to nephrocalcinosis
7. Corrected serum calcium level < 10.8 mg/dL
8. For female subjects of childbearing potential; negative urine pregnancy test and willingness to undergo additional pregnancy tests during the study
9. Willingness to use an acceptable method of contraception while participating in the study
10. Willingness to provide access to prior medical records to determine eligibility including data on imaging tests, blood chemistry, diagnosis, medication, and surgical history
11. Willingness and ability to cooperatively complete all study procedures, adhere to the visit schedule and follow the investigator's instructions, as considered by the investigator or subinvestigator

Exclusion Criteria:

1. Use of the following drugs within 14 days prior to screening: pharmacologic vitamin D metabolites or analogs, or drugs for treating TIO/ENS including oral phosphate, aluminum hydroxide antacids, acetazolamide, or thiazide diuretics
2. Medication to suppress parathyroid hormone (PTH) within 60 days prior to screening
3. Blood or blood product transfusion within 60 days prior to screening
4. Chemotherapy for TIO or other malignant tumors within 4 months prior to screening
5. History of being positive for human immunodeficiency virus antibody, hepatitis B antigen and/or hepatitis C virus antibody
6. Predisposition to infection, or history of recurrent infection or known immunodeficiency
7. Pregnant or breastfeeding at screening or intention to become pregnant during the study; for male subjects, the partner's intention to become pregnant during the study
8. Use of an investigational product or device within 4 months prior to screening, or planning to receive other investigational product before completing all assessments in this study
9. Use of therapeutic monoclonal antibodies including KRN23 within 90 days prior to screening
10. History of allergic or anaphylactic reactions to KRN23, any of the KRN23 ingredients, or any other monoclonal antibodies
11. Anyone otherwise considered unsuitable participation in the study by the investigator or subinvestigator

At the time of switching to the post-marketing study:

1. Voluntary written informed consent to participate in the post-marketing study (if aged < 20 years at the time of consent, written informed consent must be obtained from his or her legally acceptable representative as well)
2. Switching to the post-marketing study is necessary and appropriate for the subject from the viewpoint of efficacy and safety, as judged by the investigator or subinvestigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04; Primary Completion 2017-07 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
serum phosphorus concentration at each test time point | up to week 224

SECONDARY OUTCOMES:
Change from Baseline in Serum Phosphorus Level | up to week 224
Achievement Proportion of Mid-Cycle-Mean Serum Phosphorus Value (mg/dL) Exceeding the Lower Limit (2.5 mg/dL [0.81 mmol/L]) | at week 24
Achievement Proportion of End-Cycle-Mean Serum Phosphorus Value (mg/dL) Exceeding the Lower Limit (2.5 mg/dL [0.81 mmol/L]) | at week 48
Changes from baseline over time in serum Type I Collagen C-Telopeptides (CTx) | up to week 224
Changes from baseline over time in serum Procollagen 1 N-Terminal Propeptide (P1NP) | up to week 224
Changes from baseline over time in serum Bone Specific Alkaline Phosphatase (BALP) | up to week 224
Changes from baseline over time in serum Osteocalcin (OC) | up to week 224
change from baseline in FGF23 | up to week 224
change from baseline in alkaline phosphatase | up to week 224
change from baseline in 1,25(OH)2D | up to week 224
change from baseline in urine P | up to week 224
change from baseline in tubular reabsorption of phosphate | up to week 224
change from baseline in ratio of renal tubular maximum phosphate reabsorption rate to glomerular filtration rate | up to week 224
change from baseline in skeletal disease/osteomalacia through trans-iliac crest bone biopsy | up to week 224
Effect to Sit to Stand (STS) test | up to week 224
Effect to Hand Held Dynamometry (HHD) | up to week 224
Effect to Weighted Arm Lift (WAL) test | up to week 224
Effect to 6 minute walking test (6MWT) | up to week 224
Effect to patient reported outcomes | up to week 224
maximum concentration (Cmax) of KRN23 | up to week 224
area under the curve (AUC) of KRN23 | up to week 224
time to peak (tmax) of KRN23 | up to week 224

OTHER OUTCOMES:
Number and types of adverse events | up to week 224

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (2):
  - Osaka
  - Tokyo
- Seoul, South Korea